CLINICAL TRIAL: NCT04817709
Title: Development of a Patient Decision Aid for Women Considering Breast Reconstruction: User-Centered Design and Field-Testing
Brief Title: Development of a Patient Decision Aid for Women Considering Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA17-0002; NCI-2020-07838 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA17-0002 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-29; First posted 2021-03-26 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Patients view a video and read a workbook over 30 minutes about breast reconstruction surgery before their appointment. Patients also complete a questionnaire over 5-10 minutes before and after the video and after talking with the plastic surgeon. Patients' medical records are reviewed once they have made a decision about the type of reconstruction (if any).
  Interventions: Other: Educational Intervention; Other: Media Intervention; Other: Medical Chart Review; Other: Questionnaire Administration
- Arm 2: Patents receive an educational booklet about breast reconstruction surgery during appointment. Patients also complete a questionnaire over 5-10 minutes before and after talking with the plastic surgeon. Patients' medical records are reviewed once they have made a decision about the type of reconstruction (if any).
  Interventions: Other: Usual Care; Other: Medical Chart Review; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Review workbook
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Groups: Arm 1
Other: Usual Care — Receive educational materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Groups: Arm 2
Other: Media Intervention — Watch video
  Groups: Arm 1
Other: Medical Chart Review — Review of medical records
  Other Names: Chart Review
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study engages cancer survivors who have considered breast reconstruction after mastectomy in developing and pilot testing an up-to-date, understandable, meaningful patient decision aid video and workbook. Once the video and workbook are pilot-tested, a field test with new patients will then compare whether it is more feasible and useful for women considering breast reconstruction after mastectomy to view a video and workbook before their appointment or an educational booklet during their appointment. The video explains the process and types of reconstruction, the timeline for how breast reconstruction is done, and how the cost of this surgery is covered. The workbook helps patients compare your options and prepare for the appointment. The educational booklet explains the same process, types, timeline and costs, and is designed to help the patient and their surgeon compare and discuss the options together during the appointment. By comparing these two methods, researchers may learn which of these is more effective in helping patients make a decision about breast reconstruction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To design a patient decision aid video about breast reconstruction. II. To pilot test its acceptability with women. III. To field test the feasibility of delivery pre-consultation and efficacy at preparing women for their discussion with their plastic surgeon.

OUTLINE:

FOCUS GROUP: Survivors who previously considered breast reconstruction participate in a 40 to 60-minute focus group to gather feedback on currently-available patient decision aids and educational materials. The research team uses their feedback to create an initial prototype of a patient decision aid video

PILOT TEST: Survivors who previously considered breast reconstruction review the initial prototype of the patient decision aid video, then complete a questionnaire providing their feedback about the video's strengths and areas that could be improved. The research team then incorporates their feedback into the video."

FIELD TEST: Patients are randomized to 1 of 2 arms.

ARM I: Before their appointment, patients spend up to 30 minutes viewing a video and workbook. They also spend 5 to 10 minutes completing a questionnaire before and after the video and workbook, and again after their appointment. After their appointment, the research assistant reviews their medical record to confirm what decisions the patient and doctor made about breast reconstruction.

ARM II: During their appointment, patients spend up to 30 minutes reviewing the standard educational booklet about breast reconstruction. They also spend 5 to 10 minutes completing a questionnaire before and after the booklet, and again after their appointment. After their appointment, the research assistant reviews their medical record to confirm what decisions the patient and doctor made about breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Aims 1 and 2: Patients who are 6 months to 3 years post-mastectomy surgery
* Aim 3: Patients who are scheduled for their first breast reconstruction consultation with plastic surgery
* Able to speak, read, and write English

Exclusion Criteria:

* Women with cognitive or psychological impairment (e.g., depression, anxiety, severe mental illness; as documented in their medical record)
* Women for whom the video and workbook would not be appropriate due to clinical characteristics or contraindications (as determined by a provider)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are considering breast reconstruction surgery after mastectomy
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Delivery Rate | Up to 3 months prior to plastic surgery consultation
  The statistician will calculate how many women to whom the research assistant was able to deliver the video/workbook or educational materials (i.e., by sending them the URL link or scheduling time to show them the video/workbook or educational materials on an iPad at the clinic), out of the total n = 130 eligible women. The statistician will also calculate the rates of women who prefer to view the video and workbook at home or at the clinic; and of women who re-visit the video and workbook after the consultation.

SECONDARY OUTCOMES:
Breast Reconstruction Knowledge Questionnaire | Up to 3 months prior to plastic surgery consultation
  This questionnaire includes 10 true/false items assessing participants' knowledge of breast reconstruction. Items are scored such that 0% correct responses equals no knowledge and 100% correct responses equals perfect knowledge.
Preparation for Decision Making Scale | Immediately after intervention
  This questionnaire includes 11 multiple choice items assessing how well-prepared participants feel they are for making this shared medical decision with their doctors. Participants rate each item on 5-point Likert scale from 1 (Not at all) to 5 (a great deal). To calculate a total score, responses are summed and multiplied by 2 to yield the total score. Total scores range from 0 (Poorly prepared) to 100 (Excellently prepared). Alpha coefficients observed between 0.92 to 0.96. This scale discriminates between people who do/do not find the decision aid helpful (p < 0.0001). For this study, a threshold of 75 out of 100 will be considered acceptable.
Decisional Conflict Scale | Immediately before intervention, immediately after intervention, immediately after consultation
  This scale includes 16 question-items assessing participants' level of decisional conflict, defined as anxiety that blocks taking action. Participants rate each item on a Likert Scale with 5 responses from 0 (Not at All) to 4 (Extremely). Scores are summed, divided by 16, and multiplied by 25 to yield a total score of 0 (Less conflicted) to 100 (Highly conflicted). Total scores above 37.5 out of 100 are associated with delaying decisions and uncertainty about implementing their preferred treatment option; scores below 25 out of 100 are associated with making decisions and successfully implementing their preferred treatment option.
BREAST-Questionnaire (Q) | Up to 1 year prior to surgery, up to 1 year after surgery
  The BREAST-Q assesses women's self-reported ratings of their satisfaction with their breasts and associated quality of life in terms of psychosocial, sexual, and physical well-being. Participants rate 64 items from 1 (Very Dissatisfied) to 4 (Very Satisfied). Psychometric properties include a person separation index of 0.76 to 0.95, Cronbach's alphas of 0.81 to 0.96, and test-retest reproducibility of 0.73 to 0.96 Before surgery, after surgery
Type of surgery completed | Up to 1 year after surgery
  The study coordinator will abstract the type(s) of reconstructive surgery completed, including immediate versus delayed reconstruction, autologous versus implant-based reconstruction, nipple reconstruction, contralateral balancing surgery, oncoplastic tissue rearrangement, and/or no reconstruction. This questionnaire is not a validated scale and thus no scoring or psychometric properties are appropriate. Responses will be used to model potential covariate relationships with the primary and other secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reece, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org